CLINICAL TRIAL: NCT06828978
Title: Clinical and Radiographic Success Following Regenerative Pulpotomy Using Chitosan Hydrogel Versus Platelet Rich Fibrin in Mature Mandibular Molars: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Success Following Regenerative Pulpotomy Using Chitosan Hydrogel Versus Platelet Rich Fibrin in Mature Mandibular Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Perihan Adel Abdel Aziz Wafi, Resident at Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO9-1-2
Record Dates: First submitted 2024-07-17; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Regenerative Pulpotomy for Symptomatic Pulpitis of Mandibular Permanent Molars With Mature Apices

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chitosan Hydrogel after full pulpotomy (Experimental): Chitosan used as a medicament for pulpotomy as it is non-toxic biocompatible, bioadhesive, biodegradable, has wound healing ability and possesses antimicrobial activity. In addition, it encourages the odontogenic development of dental pulp stem cells.
  Interventions: Procedure: Full Pulpotomy
- Platelet Rich Fibrin after full pulpotomy (Active Comparator): Platelet-rich fibrin (PRF) is strictly autologous, biocompatible and kind toward pulp, and hence elicits minimal or nil inflammatory response when placed directly over the severed pulp.
  Interventions: Procedure: Full Pulpotomy

INTERVENTIONS:
Procedure: Full Pulpotomy — After control of bleeding in teeth allocated to the intervention group, the gel is to be placed into the pulp chamber to a level 3 mm below the cementoenamel junction (CEJ) over the root pulp stumps.

SUMMARY:
The aim of this study is to assess the clinical and radiographic success and postoperative pain in mature mandibular molars following vital pulp therapy using chitosan hydrogel versus platelet rich fibrin.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Symptomatic pulpitis in mature mandibular molars only will be involved.
* Tooth should give positive response to cold test
* Haemostasis should be achieved after full pulpotomy
* The tooth is restorable and free from advanced periodontal disease, cracks and splits.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent and will commit to follow-up period.
* Patients with mature root apices
* Patients with no internal or external resorption and no periapical lesions
* Soft tissues around the tooth are normal with no swelling or sinus tract

Exclusion Criteria:

* Patients with immature roots.
* Haemostasias after 10 minutes cannot be controlled after full pulpotomy Patients with any systemic disease that may affect normal healing.
* Patients with periapical lesions or infections.
* Pregnant females.
* Patients who could/would not participate in a 6 months follow-up.
* Patients with fistula or swelling
* Patients with necrotic pulp.
* Patients with old age.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 6 months (Postoperative)
  Using Radiographic success criteria by periapical index (Orstavik et al., 1986)

SECONDARY OUTCOMES:
Postoperative pain | 1st day up to 7th day
  Using Modified Visual Analogue Scale for pain with a straight line with one end (point 0) meaning no pain and the other end (point 10) meaning the worst pain imaginable
Tooth sensibility | 1,3,6 months (postoperative)
  Using Electric pulp test